CLINICAL TRIAL: NCT06398249
Title: Effect of Deep Breathing on Balance in Patients With Chronic Mechanical Low Back Pain
Status: Completed | Type: Observational
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Amira Mohamed Afify, Associate professor, October 6 University
Other Study IDs: P.T.REC/012/005061
Record Dates: First submitted 2024-04-16; First posted 2024-05-03 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Chronic Mechanical Low Back Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental: chronic mechanical low back pain
- control: healthy matched controls

SUMMARY:
The primary purpose of this study is to investigate the effects of deep breathing pattern on dynamic balance in patients with chronic mechanical low back pain versus healthy controls. Secondary to compare between dynamic balance control during deep versus regular breathing patterns in patients with chronic mechanical low back pain and healthy controls. Further, to detect whether pain intensity differs during balance testing applying either deep or regular breathing in patients with chronic mechanical low back pain.

DETAILED DESCRIPTION:
Diaphragm has been reported as a contributor in postural control and respiration. However, the integrated function of postural control and respiration is a complex process, especially evident during activities that increase demands on one or both functions . Previous research reports noticed that breathing pattern is altered in cases of chronic mechanical low back pain during tasks that challenges the trunk muscles function, and trunk stability . Dynamic balance control is one of the functional tasks that burdens the trunk muscles, and requires high degree of integration. Dynamic balance is disturbed in cases of chronic mechanical low back pain, and reports indicate that balance deficits extends after the painful episodes in those who have history of low back pain In patients with chronic mechanical low back pain regular respiratory movements results in greater disturbances to balance than healthy subjects .

Accordingly, in this study will attempt to emphasize the role of the deep breathing pattern during dynamic balance testing in chronic mechanical low back pain patients and matched healthy control subjects. As it is suggested that activity of the diaphragm will be focused upon through introducing deep breathing during dynamic balance testing; it is expected to enhance dynamic balance through its dual integrating its dual function of postural control and respiration.

ELIGIBILITY:
Inclusion Criteria:

* Participants in both groups should fulfill the criteria set for age and BMI ranges.
* Patients in study group should complain of pain in the lower back for a period of more than 3 months.
* Referred from an orthopedist .
* Participants in control group should haven't complained of back pain

Exclusion Criteria:

* Patients complain of radiculopathy .
* Patients complain of any other musculoskeletal disorder other than chronic mechanical low back pain .
* Any previous or current complains of pain involving other regions of the spine.
* Have history of respiratory dysfunction due to current or previous respiratory condition.
* suffer from any condition that affect balance control, including neurological, vestibular, visual or somatosensory deficits.
* use drugs that might compromise their balance control

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Their age will range between 20 and 40 years,
Study Population: Chronic low back pain patients from referrals to out patients clinics at faculty of physical therapy Cairo university. Matched healthy volunteers from students and employees of faculty of physical therapy Cairo university
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2024-02-02 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
dynamic balance testing - | At subject enrollment "single session"
  overall, mediolateral( ML), and anteroposterior(AP).
pain intensity | At subject enrollment "single session"
  visual analogue scale. A 10 cm horizontal line with one end denote "no pain" and the other end denote "severe intractable pain

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Sadat, Menofia, Egypt